CLINICAL TRIAL: NCT00988598
Title: A PHASE 1, DOUBLE-BLIND, PLACEBO-CONTROLLED, SPONSOR OPEN, RANDOMIZED, MULTIPLE DOSE STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF PF-04447943 IN MILD TO MODERATE ALZHEIMER'S DISEASE SUBJECTS ON STABLE DONEPEZIL THERAPY
Brief Title: A Brief Study To Evaluate The Safety, Tolerability, And Blood Levels Of Multiple Doses Of PF-044467943 Or Placebo In Combination With Donepezil In Subjects With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0401008
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease
Keywords: phase 1 Alzheimer's disease donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04447943 (Active Comparator)
  Interventions: Drug: PF-04447943
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04447943 — 25 mg of PF-04447943 orally every 12 hours for 7 days
  Arms: PF-04447943
Drug: Placebo — 25 mg matching placebo to PF-04447943 orally every 12 hours for 7 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety of PF-04447943 when given in combination with donepezil in subjects who have Alzheimer's Disease. The study will also evaluate the absorption and distribution of both PF-04447943 and donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have Alzheimer's dementia with a Mini Mental State Examination score between 18-26, inclusive.
* Subjects must have a reliable caregiver.
* Subjects must be on Aricept
* Memantine is allowed if subjects are on a stable dose
* Subjects must be in reasonably good health, based on medical history, physical examination, vital signs, and ECG, with no serious or unstable disease within the past 3 months.

Exclusion Criteria:

* Subjects with clinically significant heart disease cannot participate.
* Subjects with a past or current history of seizures cannot participate.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10-26 (Actual); Primary Completion 2010-07-05 (Actual); Study Completion 2010-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Glendale Adventist Medical Center, Glendale, California
  - University of Florida - Center for Clinical Trials Research, Gainesville, Florida
  - MD Clinical, Hallandale, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401008&StudyName=A%20Brief%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Blood%20Levels%20Of%20Multiple%20Doses%20Of%20PF-044467943%20Or%20Placebo%20In%20Combination%20W

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants enrolled in this study were already on prior stable donepezil therapy.
Groups:
- PF-04447943 25 mg + Donepezil: PF-04447943 25 milligram (mg) tablet orally, twice daily from Day 1 through Day 6 and once in morning on Day 7 along with donepezil 10 mg tablet orally once daily for 7 days.
- Placebo + Donepezil: Placebo matched to PF-04447943 tablet orally, twice daily from Day 1 through Day 6 and once in morning on Day 7 along with donepezil 10 mg tablet orally once daily for 7 days.
Period: Overall Study
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Started | 10 | 5
Completed | 8 | 5
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least 1 dose of study medication.
Groups:
- PF-04447943 25 mg + Donepezil: PF-04447943 25 mg tablet orally, twice daily from Day 1 through Day 6 and once in morning on Day 7 along with donepezil 10 mg tablet orally once daily for 7 days.
- Total: Total of all reporting groups
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (5.6) | 69.8 (5.8) | 69.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vital Signs Abnormalities of Potential Clinical Concern
Description: Criteria for vital signs abnormalities of potential concern included: supine/standing systolic blood pressure (BP) (less than [<] 90 millimeter of mercury [mmHg], maximum [max] decrease and increase of greater than or equal to [>=] 30 mmHg from baseline); diastolic BP (<50 mmHg, maximum decrease and increase of >=20 mmHg from baseline); supine pulse rate <40 beats per minute [bpm] or greater than [>]120 bpm); standing pulse rate <40 bpm or >140 bpm. Baseline is defined as the last pre-dose (PF-04447943) recording at Day 0.
Time Frame: Baseline up to Day 10
Population: Safety analysis set included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
participants
  Supine Systolic BP (<90 mmHg) | 0 | 0
  Standing Systolic BP (<90 mmHg) | 0 | 0
  Supine Diastolic BP (<50 mmHg) | 0 | 0
  Standing Diastolic BP (<50 mmHg) | 0 | 0
  Max Increase in Supine Systolic BP (>=30 mmHg) | 0 | 2
  Max Increase in Standing Systolic BP (>=30 mmHg) | 0 | 2
  Max Increase in Supine Diastolic BP (>=20 mmHg) | 1 | 1
  Max Increase in Standing Diastolic BP (>=20 mmHg) | 0 | 1
  Max Decrease in Supine Systolic BP (>=30 mmHg) | 2 | 1
  Max Decrease in Standing Systolic BP (>=30 mmHg) | 2 | 1
  Max Decrease in Supine Diastolic BP (>=20 mmHg) | 0 | 1
  Max Decrease in Standing Diastolic BP (>=20 mmHg) | 0 | 0
  Supine Pulse Rate (<40 bpm) | 0 | 0
  Supine Pulse Rate (>120 bpm) | 0 | 0
  Standing Pulse Rate (<40 bpm) | 0 | 0
  Standing Pulse Rate (>140 bpm) | 0 | 0

2. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities of Potential Clinical Concern
Description: Criteria for ECG abnormalities of potential clinical concern included: PR interval (>=300 milliseconds [msec], >= 25 percent [%] increase when baseline >200 msec or increase >=50% when baseline less than or equal to [<=] 200 msec); QRS interval (>=200 msec, >= 25% increase when baseline >100 msec or increase >=50% when baseline <=100 msec); QT corrected using Fridericia's formula (QTcF) (>=500 msec, maximum increase between >=30 to <60 msec and >=60 msec). Baseline is defined as the last pre-dose (PF-04447943) recording at Day 0.
Time Frame: Baseline up to Day 10
Population: Safety analysis set included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
participants
  Maximum PR Interval (>=300 msec) | 0 | 0
  Maximum PR Interval Increase (>=25/50%) | 0 | 0
  Maximum QRS Interval (>=200 msec) | 0 | 0
  Maximum QRS Interval Increase (>=25/50%) | 0 | 0
  Maximum QTcF Interval (>=500 msec) | 0 | 0
  Maximum QTcF Interval Increase(Change >=30 to <60) | 2 | 1
  Maximum QTcF Interval Increase (Change >=60) | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit (<0.8*lower limit of normal [LLN]); red blood cell count (<0.8*LLN); platelets (<0.5*LLN or >1.75* upper limit of normal [ULN]); leucocytes (<0.6*LLN or >1.5*ULN); lymphocytes, total neutrophils (<0.8*LLN or >1.2*ULN); basophils, eosinophils, monocytes (>1.2*ULN); total bilirubin (>1.5* ULN); aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase (>3*ULN); creatinine, blood urea nitrogen (>1.3*ULN); glucose (<0.6*LLN or >1.5*ULN); uric acid (>1.2*ULN); sodium (<0.95*LLN or 1.05*ULN); potassium, calcium, chloride, bicarbonate (<0.9*LLN or 1.1*ULN); albumin, total protein (<0.8*LLN or 1.2*ULN); urine analysis. Total number of participants with any laboratory abnormalities was reported.
Time Frame: Baseline up to Day 10
Population: Safety analysis set included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
participants | 4 | 4

4. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 10 after last dose that were absent before treatment or that worsened relative to pretreatment state. Any abnormalities related to physical and neurological findings, laboratory tests, vital signs and ECG were reported as adverse events. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to Day 10
Population: Safety analysis set included all participants who had received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
participants
  AEs | 6 | 0
  SAEs | 0 | 0

5. Secondary Outcome: Plasma Concentrations of PF-04447943
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours after morning dose of PF-04447943 on Day 1, Day 7
Population: Pharmacokinetic (PK) concentration analysis set included all randomized participants who had received at least one dose of PF-04447943 and had at least 1 evaluable PF-04447943 concentration. Here, 'number analyzed, n' signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04447943 25 mg + Donepezil
Number analyzed (Participants) | 10
nanogram per milliliter (ng/mL)
  Day 1: 0 hours | 0.01050 (0.033204)
  Day 1: 0.5 hours | 179.6 (127.67)
  Day 1: 1 hour | 296.7 (83.312)
  Day 1: 3 hours | 225.9 (46.905)
  Day 1: 8 hours | 91.76 (30.400)
  Day 1: 12 hours | 51.99 (21.018)
  Day 7: 0 hours: number analyzed (Participants) | 8
  Day 7: 0 hours | 73.49 (28.023)
  Day 7: 0.5 hours: number analyzed (Participants) | 8
  Day 7: 0.5 hours | 340.4 (168.41)
  Day 7: 1 hour: number analyzed (Participants) | 8
  Day 7: 1 hour | 353.6 (112.63)
  Day 7: 3 hours: number analyzed (Participants) | 8
  Day 7: 3 hours | 284.0 (83.881)
  Day 7: 8 hours: number analyzed (Participants) | 8
  Day 7: 8 hours | 124.8 (49.247)
  Day 7: 12 hours: number analyzed (Participants) | 8
  Day 7: 12 hours | 69.08 (28.483)

6. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-04447943
Description: Area under the plasma concentration time-curve from time zero to end of dosing interval (tau), where dosing interval is 12 hours.
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours after morning dose of PF-04447943 on Day 1, Day 7
Population: PK analysis set included all randomized participants who had received at least one dose of PF-04447943 and had at least 1 of the PK parameters of interest for PF-04447943. Here, 'n' signifies those participants who were evaluable at specified time point.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-04447943 25 mg + Donepezil
Number analyzed (Participants) | 10
nanogram*hour per milliliter (ng*hr/mL)
  Day 1 | 1657 (391.88)
  Day 7: number analyzed (Participants) | 8
  Day 7 | 2140 (688.96)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04447943
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours after morning dose of PF-04447943 on Day 1, Day 7
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04447943 25 mg + Donepezil
Number analyzed (Participants) | 10
ng/mL
  Day 1 | 303.8 (66.655)
  Day 7: number analyzed (Participants) | 8
  Day 7 | 390.9 (109.31)

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04447943
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours after morning dose of PF-04447943 on Day 1, Day 7
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04447943 25 mg + Donepezil
Number analyzed (Participants) | 10
hours
  Day 1 | 1.00 [1.00 to 3.00]
  Day 7: number analyzed (Participants) | 8
  Day 7 | 0.767 [0.500 to 3.00]

9. Secondary Outcome: Plasma Concentrations of Donepezil
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours post donepezil administration on Day 0(Baseline), Day 7
Population: PK concentration analysis set included all randomized participants who had received donepezil and had at least 1 evaluable donepezil concentration. Here, 'n' signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
ng/mL
  Day 0: 0 hours | 29.30 (22.982) | 19.10 (10.562)
  Day 0: 0.5 hours | 29.93 (22.874) | 23.92 (16.478)
  Day 0: 1 hour | 41.08 (20.592) | 36.18 (9.6916)
  Day 0: 3 hours | 54.09 (28.122) | 41.56 (11.088)
  Day 0: 8 hours | 42.15 (24.360) | 30.92 (11.339)
  Day 0: 12 hours: number analyzed (Participants) | 9 | 5
  Day 0: 12 hours | 34.04 (20.659) | 28.02 (11.308)
  Day 7: 0 hours: number analyzed (Participants) | 8 | 5
  Day 7: 0 hours | 34.94 (22.579) | 33.86 (3.7031)
  Day 7: 0.5 hours: number analyzed (Participants) | 8 | 5
  Day 7: 0.5 hours | 39.56 (26.766) | 35.82 (3.8226)
  Day 7: 1 hour: number analyzed (Participants) | 8 | 5
  Day 7: 1 hour | 47.29 (30.726) | 45.04 (12.347)
  Day 7: 3 hours: number analyzed (Participants) | 8 | 5
  Day 7: 3 hours | 58.15 (30.916) | 56.36 (5.6783)
  Day 7: 8 hours: number analyzed (Participants) | 8 | 5
  Day 7: 8 hours | 46.90 (23.802) | 45.42 (4.4404)
  Day 7: 12 hours: number analyzed (Participants) | 8 | 5
  Day 7: 12 hours | 42.83 (23.299) | 41.78 (4.7505)

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Donepezil
Description: Area under the plasma concentration time-curve from time zero to end of dosing interval (tau), where dosing interval is 24 hours.
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours post donepezil administration on Day 0(Baseline), Day 7
Population: PK analysis set included all randomized participants who had received donepezil and had at least 1 of the PK parameters of interest of donepezil. Here, 'n' signifies those participants who were evaluable at specified time point.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
ng*hr/mL
  Day 0 | 426.8 (256.08) | 380.6 (127.02)
  Day 7: number analyzed (Participants) | 8 | 5
  Day 7 | 513.4 (314.66) | 565.2 (40.402)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Donepezil
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours post donepezil administration on Day 0(Baseline), Day 7
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
ng/mL
  Day 0 | 47.60 (27.600) | 42.48 (8.1522)
  Day 7: number analyzed (Participants) | 8 | 5
  Day 7 | 52.88 (30.177) | 59.61 (4.6404)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Donepezil
Time Frame: 0 hours (pre-dose), 0.5, 1, 3, 8, 12 hours post donepezil administration on Day 0(Baseline), Day 7
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Number analyzed (Participants) | 10 | 5
hours
  Day 0 | 3.00 [1.00 to 3.00] | 3.00 [1.00 to 3.02]
  Day 7: number analyzed (Participants) | 8 | 5
  Day 7 | 3.00 [1.00 to 8.00] | 3.00 [1.00 to 3.00]

ADVERSE EVENTS:
Arm/Group | PF-04447943 25 mg + Donepezil | Placebo + Donepezil
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 6/10 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04447943 25 mg + Donepezil (N=10) | Placebo + Donepezil (N=5)
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.